CLINICAL TRIAL: NCT02082262
Title: AGN-229666 Ophthalmic Solution for the Treatment of Seasonal or Perennial Allergic Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 229666-005
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Results first posted 2015-10-08 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Conjunctivitis, Allergic
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AGN-229666 (Experimental): One to two drops of AGN-229666 twice daily in each eye for 10 weeks.
  Interventions: Drug: AGN-229666

INTERVENTIONS:
Drug: AGN-229666 — One to two drops of AGN-229666 twice daily in each eye for 10 weeks.

SUMMARY:
This study will evaluate the safety and efficacy of AGN-229666 for the treatment of seasonal or perennial allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients living in Japan with allergic conjunctivitis with itching and redness
* Able and willing to discontinue wearing any contact lenses during the study period.

Exclusion Criteria:

* Eye surgical intervention and/or a history of refractive surgery within 6 months
* History of retinal detachment, diabetic retinopathy, or progressive retinal disease
* Presence of active eye infection (bacterial, viral, or fungal)
* History of an eye herpetic infection
* Use of corticosteroids within 6 months or anticipated use during the study.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AGN-229666
Started | 140
Completed | 89
Not Completed | 51
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 48

BASELINE CHARACTERISTICS:
Arm/Group | AGN-229666
Number analyzed (Participants) | 140
Age, Customized [Number; unit: Participants]
  ≥ 10 to < 20 years | 38
  ≥ 20 to < 40 years | 44
  ≥ 40 years | 58
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 58

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline In Ocular Itching Frequency Score Using a 6-point Scale
Description: Ocular itching frequency is assessed on a 6-poing scale, where 0 = did not occur, 1 = once in 3 days, 2 = twice in 3 days, 3 = once every day, 4 = 2 or more times every day, and 5 = virtually all the time over the past 3 days. Ocular itching frequency is evaluated over the 3 days prior to the visit. A negative number change from baseline indicates an improvement and a positive number change from baseline indicates a worsening.
Time Frame: Baseline, Day 70
Population: Modified Intent-to-Treat: all enrolled patients with at least one follow-up ocular itching frequency score
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | AGN-229666
Number analyzed (Participants) | 140
Scores on a Scale
  Baseline | 4.4 (0.49)
  Change from Baseline at Day 70 (N=110) | -3.4 (1.51)

ADVERSE EVENTS:
Arm/Group | AGN-229666
Serious Adverse Events (participants affected / at risk) | 0/140
Other Adverse Events (participants affected / at risk) | 96/140
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-229666 (N=140)
Conjunctival Hyperaemia (Eye disorders) | 48
Eye Pruritus (Eye disorders) | 28
Somnolence (Nervous system disorders) | 26
Eye Discharge (Eye disorders) | 14
Instillation Site Irritation (General disorders) | 12
Ciliary Hyperaemia (Eye disorders) | 11
Eyelid Oedema (Eye disorders) | 9
Blepharitis (Eye disorders) | 8
Conjunctivitis (Eye disorders) | 8
Conjunctival Oedema (Eye disorders) | 7
Nasopharyngitis (Infections and infestations) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.